CLINICAL TRIAL: NCT05086133
Title: The Effect of cTBS on First-episode Drug Naive Patients With Schizophrenia
Brief Title: cTBS on First-episode Drug Naive Patients With Schizophrenia
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Active, not recruiting
Sponsor: Central South University (Other)
Collaborators: Shanghai Mental Health Center (Other)
Responsible Party: Principal Investigator, Renrong Wu, Professor, Central South University
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: WU2021TBS
Record Dates: First submitted 2021-09-23; First posted 2021-10-20 (Actual); Last update posted 2022-11-17 (Actual); Status verified 2022-11

CONDITIONS: Schizophrenia
MeSH Terms: conditions — Schizophrenia | interventions — Transcranial Magnetic Stimulation

STUDY DESIGN:
Intervention Model Description: 1 group for intervention and 1 group for sham stimulation
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Masking Description: The participants will be randomized into experimental group or sham group by a predetermined randomization table. The participants, care provider, investigators and outcomes assessor will be blind to the grouping. The physician who perform the TMS intervention is not blind to the grouping.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- cTBS stimulation (Experimental): The participants randomized into experimental group will receive cTBS stimulation of left M1 area for 5 times a day, with 1h interval between two stimulations, and for 5 continuous days.
  Interventions: Device: transcranial magnetic stimulation
- Sham stimulation (Sham Comparator): The participants randomized into experimental group will receive sham stimulation of left M1 area for 5 times a day, with 1h interval between two stimulations, and for 5 continuous days.
  Interventions: Device: sham stimulation

INTERVENTIONS:
Device: transcranial magnetic stimulation — transcranial magnetic stimulation with continuous theta burst pattern, 90% RMT, 50Hz within train and 5Hz train for 200 train and 40 second in total.
  Arms: cTBS stimulation
Device: sham stimulation — TMS coil vertical to the brain surface, with same protocol as cTBS
  Arms: Sham stimulation

SUMMARY:
cTBS is a promising novel intervention, which have strong potentials on moderating disease syndrome, suck as verbal hallucination, and cognitive deficits in schizophrenia, as it has been proved for the treatment of depression.

Therefore, the investigators designed this randomized controlled clinical trial to evaluate the efficacy and safety of cTBS on prevention and treatment for cognitive deficiency, psychotic syndrome and metabolic side-effects in drug-naive first episode individual with schizophrenia.

DETAILED DESCRIPTION:
cTBS is a promising novel intervention, which have strong potentials on moderating disease syndrome, suck as verbal hallucination, and cognitive deficits in schizophrenia, as it has been proved for the treatment of depression.

Therefore, the investigators designed this randomized controlled clinical trial to evaluate the efficacy and safety of cTBS on prevention and treatment for cognitive deficiency, psychotic syndrome and metabolic side-effects in drug-naive first episode individual with schizophrenia.

ELIGIBILITY:
Inclusion Criteria:

* Patients diagnosed with schizophrenia in accordance with DSM-5
* The course of the disease less then 2 years
* Accepting antipsychotics treatment for less then 2 months

Exclusion Criteria:

* Diagnosed with other mental disease in accordance with DSM-5
* Comorbid with other severe physiological disease
* Used antipsychotic, antidepressants, mood stabilizer, or other psychoactive substances before
* Drug or alcohol abuse
* Pregnant or lactating Contraindication to rTMS

Ages: 18 Years to 40 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 44 (Actual)
Dates: Start 2021-11-20 (Actual); Primary Completion 2022-11-15 (Actual); Study Completion 2023-06-01 (Estimated)

PRIMARY OUTCOMES:
Three-Factor Eating Questionnaire | Change from Baseline to 6days and 36days
  min value 21, max value 84. The higher scores mean more unhealthy eating behavior.
MCCB | Change from Baseline to 6days and 36days
  The MATRICS™ Consensus Cognitive Battery
The positive and negative syndrome scale | Change from Baseline to 6days and 36days
  min score 30, max score 210. The higher score means more severe symptoms.
BMI | Change from Baseline to 6days and 36days
  body mass index

SECONDARY OUTCOMES:
Resting EEG | Change from Baseline to 6days and 36days
  resting EEG (electroencephalogram) with eyes opened, eye closed and natural stimulation. The reEEG power spectra, functional connection will be calculated.
fasting glucose | Change from Baseline to 6days and 36days
  in mmol/l
Triglyceride | Change from Baseline to 6days and 36days
  in mmol/l
Total Cholesterol | Change from Baseline to 6days and 36days
  in mmol/l
Low Density Lipoprotein | Change from Baseline to 6days and 36days
  in mmol/l
High Density Lipoprotein | Change from Baseline to 6days and 36days
  in mmol/l

CONTACTS AND LOCATIONS:
Locations (1):
- Central South University, Changsha, Hunan, China

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Kang D, Song C, Peng X, Yu G, Yang Y, Chen C, Long Y, Shao P, Wu R. The effect of continuous theta burst stimulation on antipsychotic-induced weight gain in first-episode drug-naive individuals with schizophrenia: a double-blind, randomized, sham-controlled feasibility trial. Transl Psychiatry. 2024 Jan 25;14(1):61. doi: 10.1038/s41398-024-02770-w. PMID 38272892
- [Derived] Kang D, Zhang Y, Wu G, Song C, Peng X, Long Y, Yu G, Tang H, Gui Y, Wang Q, Yuan T, Wu R. The Effect of Accelerated Continuous Theta Burst Stimulation on Weight Loss in Overweight Individuals With Schizophrenia: A Double-Blind, Randomized, Sham-Controlled Clinical Trial. Schizophr Bull. 2024 Apr 30;50(3):589-599. doi: 10.1093/schbul/sbad144. PMID 37921353